CLINICAL TRIAL: NCT01939353
Title: An Exploratory, Single-Blind Pilot Trial of Flexible Doses of the Triple Reuptake Inhibitor EB-1020 SR in the Treatment of Adult Males With Attention-Deficit Hyperactivity Disorder
Brief Title: Study of Flexible Doses of the Triple Reuptake Inhibitor EB-1020 Sustained Release (SR) in the Treatment of Adult Males With Attention-Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EB-1020-SR-ADHD-201
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Adult ADHD
Keywords: Adult ADHD; centanafadine sustained release
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Masking Description: This was a single-blind trial in which participants were blinded to investigational product throughout the trial. Participants were not informed of the exact timing of CTN SR versus placebo treatment, in order to maintain the blinded nature of the placebo treatment and reduce potential placebo effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Centanafadine SR 100-500 mg (Experimental): Following a 1-week SB placebo run-in treatment, participants with <30% improvement and ≥28 total score on Adult ADHD-RS-IV scale score received centanafadine (CTN) 100 mg, sustained release (SR) tablet, once daily (1 tablet in the morning) on Days 1 and 2, followed by 200 mg, SR tablets, twice daily (1 tablet in the morning and 1 tablet 5 hours later) on Days 3 and 4, followed by 300 mg, SR tablets, twice daily (2 tablets in the morning and 1 tablet 5 hours later) on Days 5, 6, and 7. After 1 week of treatment, CTN doses were maintained or titrated in 100-mg increments up to the maximum of 500 mg daily or reduced based on the safety and tolerability, as judged by the investigator at Weeks 2, 3 and 4.
  Interventions: Drug: CTN SR; Drug: Placebo

INTERVENTIONS:
Drug: CTN SR — CTN SR tablets
  Other Names: EB-1020 SR
Drug: Placebo — CTN SR-matching placebo tablets

SUMMARY:
This was a Phase 2 exploratory study to evaluate the efficacy and safety of EB-1020 SR (centanafadine sustained release [CTN SR]) in treating participants who met Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) diagnostic criteria for Attention-Deficit Hyperactivity Disorder (ADHD) on the Mini International Neuropsychiatric Interview Plus, Version 6.0 (M.I.N.I.-Plus). Evaluations included determining an effectiveness signal for ADHD and related symptoms and exploring dosing, tolerability, onset of action, and duration of effect. Dose-response/tolerability relationships with CTN SR were also explored. The 1-week placebo run-in [single-blind (SB)] was also used for informal safety comparison purposes.

DETAILED DESCRIPTION:
This Phase 2, flexible-dosage, single-blind exploratory study of CTN SR in adult male participants with ADHD consisted of a 1-week placebo run-in (SB), 4 weeks of treatment with CTN SR, and 2 weeks of follow-up. At the placebo run-in, participants must have had a score of greater than or equal to 28 on the Adult Attention-Deficit Hyperactivity Disorder Rating Scale Version IV (ADHD-RS-IV) to be eligible to continue participation in the study.

At the end of single-blind placebo run-in treatment (that is, beginning of CTN SR treatment), the ADHD-RS-IV with adult prompts was re-administered. Participants who showed an improvement greater than or equal to 30% over baseline values or who had a score of less than 28 on the ADHD-RS-IV were withdrawn from the study prior to receiving any active drug. Those who showed less than 30% improvement from the placebo run-in to the beginning of CTN SR treatment continued the study. The consent form was phrased such that participants were not informed of the exact timing of CTN SR versus placebo treatment in order to maintain the blinded nature of the placebo treatment and reduce potential placebo effects. Dosing was flexible, with a target maximum dosage of 500 milligrams (mg) daily in divided doses (morning and afternoon, approximately 5 hours later) to be achieved if possible during Week 2 of CTN SR treatment. The participants took a starting dose of 100 mg of CTN SR daily; the dose was titrated in 100 mg increments up to the maximum dosage of 500 mg daily. The treating physician escalated the dose to the maximum dose if participants had not achieved remission of ADHD in his/her judgment, and CTN SR was still well tolerated. If in the physician's judgment the participant could not tolerate further dose escalation, or was not tolerating the current dose well, the dose was maintained or reduced, with the goal of re-assessing dose and response at the subsequent visit for a possible increase in dose, until study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Participants had to be able to understand the nature of the study, agree to comply with the prescribed dosage regimens, report for regularly scheduled office visits, and communicate to study personnel about adverse events and concomitant medication use.
2. Participants must have met DSM-IV-TR diagnostic criteria for ADHD (Combined, Predominantly Inattentive or Predominantly Hyperactive-Impulsive Types) on the M.I.N.I.-Plus.
3. Participants must have had an ADHD-RS-IV score of greater than or equal to 28 at the placebo run-in baseline and CTN SR treatment baseline.
4. Participants must have had a Clinical Global Impression of Severity (ADHD version) score of greater than or equal to 4.
5. Participants must be able to read well enough to understand the informed consent form and other participant materials.
6. Participants must have been able to be reliably rated on the psychiatric scales required by the protocol based on investigator's judgment.
7. Participants must have been able to read and understand English.
8. Participants must have had a body mass index of approximately 18 to 35 kilograms/meter squared.
9. Sexually active, fertile males must have used effective birth control if their partners were women of childbearing potential. Women of childbearing potential (if a partner of a male participant) included any female who had experienced menarche and who had not undergone successful surgical sterilization or women on hormone replacement therapy with documented serum follicle stimulating hormone level greater than 35 milli-international units/milliliter. Even women who were using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or were practicing abstinence or where the partner was sterile (for example, vasectomy), should have been considered to be of childbearing potential.

Exclusion Criteria:

1. Participant had a DSM-IV-TR diagnosis of ADHD not otherwise specified.
2. Participants rated as having a greater than or equal to 30% improvement in ADHD symptoms or a score of less than 28 on the ADHD-RS-IV after Week 1 (placebo run-in). Such participants were withdrawn from the study prior to receiving any active drug.
3. Participant had a current or lifetime history of bipolar disorder or any psychotic disorder as established by M.I.N.I.-Plus.
4. Participant had a current history (past 90 days) of major depression, generalized anxiety disorder, obsessive-compulsive disorder, panic disorder or post-traumatic stress disorder as established by the M.I.N.I.-Plus.
5. History in the past 20 years of electroconvulsive therapy or lifetime history of vagal nerve stimulation or deep brain stimulation for the treatment of depression.
6. Participants with a history of drug or alcohol use disorders (abuse or dependence) must have been free of the diagnosis and of substance use for at least 6 months prior to the Screening visit.
7. Participant had a history of epilepsy, seizures, syncope, unexplained blackout spell(s), head trauma with clinically significant loss of consciousness or noninfantile febrile seizures.
8. Participant had a currently active medical condition (other than ADHD) that, in the opinion of the investigator, could have interfered with the ability of the participant to participate in the study safely.
9. Participant had a history of clinically significant, diagnosed cardiovascular disease of any kind, including uncontrolled hypertension. Participant had newly diagnosed cardiovascular disease of any kind in the investigator's judgment.
10. The participant had an intelligence quotient less than 80.
11. In the opinion of the investigator, the participant had not derived significant therapeutic benefit from 2 or more ADHD therapies given with an adequate dose and duration in adulthood (age 18 or older); that is, 1 failed course of treatment was acceptable, but 2 failed courses of treatment were not acceptable.
12. Participant taking medication specifically for treatment of ADHD symptoms (for example, stimulants, atomoxetine, tricyclic antidepressants, bupropion, modafinil) must have been off stimulants for 2 weeks and off nonstimulant ADHD therapies for 3 weeks prior to the placebo run-in visit and must have returned to the baseline level of ADHD symptoms in the opinion of the investigator. Participants must not have had evidence of a discontinuation or withdrawal reaction.
13. Participant was currently taking any antidepressant medication for any condition.
14. Participant was currently taking antipsychotic medication or an anticonvulsant medication (for example, phenytoin, carbamazepine, lamotrigine, or valproic acid) at anticonvulsant doses.
15. Participant had a known history of allergy to CTN.
16. Participant was unwilling to refrain from taking medications that may have interfered with the assessment of cognitive function and the assessment of sleep. Examples included benzodiazepines, sedating antihistamines, zolpidem, eszopiclone, and zaleplon. Herbal preparations with effects on the central nervous system also were prohibited throughout the study (for example, St. John's Wort or melatonin).
17. Participant had a history of sleep problems in the last 3 months.
18. Participant was unwilling to refrain from taking more than 1 unit of alcohol within 24 hours of the investigational center visits.
19. Participant was unwilling to restrict caffeine to no more than 500 mg/day (5 cups of coffee).
20. Participant was actively using any drugs with potential for abuse (for example, marijuana, cocaine, amphetamines).
21. Participant reported passive or active suicidal ideation or intent.
22. Participant was concurrently participating in another clinical research study or investigational drug study or had participated in such a study within the past 1 month.
23. Participant was at high risk of nonadherence to investigational product and the protocol regimen in the investigator's opinion.
24. Participant could not have begun psychotherapy during the study, but may have continued therapy at the same intensity and frequency, if begun at least 3 months prior to placebo run-in.

Exclusion Criteria, Physical and Laboratory Test Findings

1. Participants who had a positive urine drug screen, which could not be explained by prescribed medications. The urine drug screen may have been repeated based on investigator judgment.
2. Participants with clinically significantly abnormal thyroid-stimulating hormone or a positive result on a standard hepatitis-screening panel or human immunodeficiency virus screen. Note: Adequate thyroid replacement for a previously diagnosed thyroid deficiency, which had been stable for 3 months or more, was acceptable.
3. Participants with clinically significant laboratory abnormalities or with clinical laboratory values of potential clinical concern.
4. Diastolic blood pressure greater than 85 millimeters of mercury (mmHg) at placebo run-in.
5. Systolic blood pressure greater than 135 mmHg at placebo run-in.
6. Participant had a QT interval of greater than 450 milliseconds on 2 or more electrocardiogram tracings taken within 15 minutes, assessed with the participant in a supine position for 3 minutes.

Other Exclusion Criteria

1. Prisoners or participants who were involuntarily incarcerated.
2. Participants who had a compulsory detainment for treatment of either a psychiatric or a physical illness.
3. Participants who planned to have elective surgeries during the course of the study.
4. Participants with a history of antidepressant-induced hypomania or dysphoria.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bradenton, Florida
  - Maitland, Florida
  - Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- Available data/document: Poster Abstracts — https://apsard.org/wp-content/uploads/2016/11/Poster-Abstracts-Compiled1.pdf — Poster number 25

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 03 October 2013 to 20 February 2014.
Pre-assignment Details: A total of 45 male participants diagnosed with attention-deficit hyperactivity disorder (ADHD) were enrolled at Baseline-1 in a 1-week single-blind (SB) placebo run-in treatment to receive placebo from Baseline-1 to Baseline-2. At Baseline-2, remaining 41 out of 45 participants who had <30% improvement and ≥28 total score on Adult ADHD-RS-IV scale score received centanafadine (CTN) sustained release (SR) 100-500 mg, tablets from Week 1 to Week 4.
Groups:
- Centanafadine SR 100-500 mg: Following a 1-week SB placebo run-in treatment, participants with <30% improvement and ≥28 total score on Adult ADHD-RS-IV scale score received CTN 100 mg, SR tablet, once daily (1 tablet in the morning) on Days 1 and 2, followed by 200 mg, SR tablets, twice daily (1 tablet in the morning and 1 tablet 5 hours later) on Days 3 and 4, followed by 300 mg, SR tablets, twice daily (2 tablets in the morning and 1 tablet 5 hours later) on Days 5, 6, and 7. After 1 week of treatment, CTN doses were maintained or titrated in 100-mg increments up to the maximum of 500 mg daily or reduced based on the safety and tolerability, as judged by the investigator at Weeks 2, 3 and 4.
Period: Placebo Run-in (1 Week)
Arm/Group | Centanafadine SR 100-500 mg
Started | 45
Completed | 41
Not Completed | 4
Not completed — Withdrew Consent | 3
Not completed — Lost to Follow-up | 1
Period: CTN SR Treatment Phase (4 Weeks)
Arm/Group | Centanafadine SR 100-500 mg
Started | 41
Completed | 37
Not Completed | 4
Not completed — Treatment Emergent Adverse Event (TEAE)/Serious Adverse Event (SAE) | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of CTN SR (not placebo) as indicated in the treatment regimen.
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.71 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 37
  Race: Black or African American | 03
  Race: Asian | 01
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 04
  Ethnicity: Not Hispanic or Latino | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline-2 in ADHD Symptoms to Week 4 as Assessed by the Adult Attention-Deficit Hyperactivity Disorder Rating Scale (AD HD-RS-IV)
Description: The ADHD-RS-IV consists of 18 items with first 9 items assessing inattentive symptoms and the last 9 items assessing hyperactive-impulsive symptoms scored on a 4-point Likert-type severity scale with 0 (none), 1 (mild), 2 (moderate), and 3 (severe) with a total score ranging from 0 to 54. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 4
Population: Per-protocol Population included all participants who met inclusion/exclusion criteria and completed the trial (4 weeks of drug treatment with evaluable data after Week 4) without major protocol violations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  Baseline-2 | 38.70 (6.19)
  Change from Baseline-2 at Week 4 | -21.41 (10.74)

2. Secondary Outcome: Change From Baseline-2 in ADHD Symptoms as Assessed by the Adult ADHD-RS-IV
Description: as for outcome 1
Time Frame: Baseline-2, Weeks 1, 2, 3, and 6 (Follow-up Visit)
Population: Per-protocol Population included all participants who met inclusion/exclusion criteria and completed the trial (4 weeks of drug treatment with evaluable data after Week 4) without major protocol violations. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  Baseline-2 | 38.70 (6.19)
  Change from Baseline-2 at Treatment Week 1 | -11.14 (8.64)
  Change from Baseline-2 at Treatment Week 2 | -16.14 (11.08)
  Change from Baseline-2 at Treatment Week 3 | -20.86 (11.11)
  Change from Baseline-2 at Week 6 (Follow-up Visit): number analyzed (Participants) | 36
  Change from Baseline-2 at Week 6 (Follow-up Visit) | -11.53 (8.78)

3. Secondary Outcome: Change From Baseline-2 to Week 4 on the Behavior Rating Inventory of Executive Function, Adult Version (BRIEF-A) Scale
Description: BRIEF-A is a standardized self-administered scale that captures an adult's executive functions or self-regulation in their everyday environment, composed of 75 items within 9 nonoverlapping derived clinical scales and measures various aspects of executive functioning, including the following: inhibit, self-monitor shift, emotional control, initiate, working memory, plan/organize, monitor, and organization of materials. Items are rated 1=never, 2=sometimes, and 3=often; total raw scale score ranges from 75-225, higher total scores=more problems with executive functioning. Raw scale scores are used to generate T-scores. Total T-scores range from 30 to 90, with broader composite indexes including Behavioral Regulation Index(BRI) and Metacognition Index(Ml). These indexes form overall summary score, the Global Executive Composite(GEC). Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR. A negative change from Baseline indicates improvement.
Time Frame: Baseline-2 and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  RAW Score: BRI at Baseline-2 | 57.11 (10.96)
  RAW Score: Change from Baseline-2 in BRI at Week 4 | -8.38 (9.42)
  RAW Score: MI at Baseline-2 | 88.08 (13.46)
  RAW Score: Change from Baseline-2 in MI at Week 4 | -13.70 (15.69)
  RAW Score: GEC at Baseline-2 | 145.19 (22.27)
  RAW Score: Change from Baseline-2 in GEC at Week 4 | -22.08 (24.54)
  T-Score: BRI at Baseline-2 | 65.62 (11.99)
  T-Score: Change from Baseline-2 in BRI at Week 4 | -8.93 (10.07)
  T-Score: MI at Baseline-2 | 74.26 (10.71)
  T-Score: Change from Baseline-2 in MI at Week 4 | -10.83 (12.37)
  T-Score: GEC at Baseline-2 | 71.86 (11.43)
  T-Score: Change from Baseline-2 in GEC at Week 4 | -10.86 (12.04)

4. Secondary Outcome: Percentage of Participants Who Are Responders for ADHD Symptoms as Measured by the ADHD-RS-IV
Description: Responders are defined as participants with ≥30% improvement in ADHD symptoms compared with Baseline-2, as measured by the ADHD-RS-IV. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR.
Time Frame: Baseline-2, Weeks 1, 2, 3, and 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
percentage of participants
  Week 1 | 35.14
  Week 2 | 62.16
  Week 3 | 75.68
  Week 4 | 81.08

5. Secondary Outcome: Percentage of Participants Who Are High Responders for ADHD Symptoms as Measured by the ADHD-RS-IV
Description: High responders are defined as participants with ≥50% improvement in ADHD symptoms compared with Baseline-2, as measured by the ADHD-RS-IV. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR.
Time Frame: Baseline-2, Weeks 1, 2, 3, and 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
percentage of participants
  Week 1 | 16.22
  Week 2 | 43.24
  Week 3 | 62.16
  Week 4 | 62.16

6. Secondary Outcome: Change From Baseline-2 on the Inattentiveness and Hyperactivity/Impulsivity Subscales of ADHD-RS-IV
Description: The ADHD-RS-IV consists of 18 items with first 9 items assessing inattentive symptoms and the last 9 items assessing hyperactive-impulsive symptoms scored on a 4-point Likert-type severity scale with 0=none, 1=mild, 2=moderate, and 3=severe, with a total score ranging from 0 to 54. Inattention and hyperactivity/impulsivity subscales consist of 9 items each, for total subscale scores ranging from 0 to 27. Higher scores are indicative of more severe symptoms. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR. A negative change from Baseline indicates improvement.
Time Frame: Baseline-2, Weeks 1, 2, 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  Inattention Symptoms at Baseline-2 | 22.81 (2.55)
  Change from Baseline-2 in Inattention Symptoms at Week 1 | -6.32 (4.99)
  Change from Baseline-2 in Inattention Symptoms at Week 2 | -9.76 (6.40)
  Change from Baseline-2 in Inattention Symptoms at Week 3 | -12.16 (6.61)
  Change from Baseline-2 in Inattention Symptoms at Week 4 | -12.41 (6.66)
  Hyperactive/Impulsive Symptoms at Baseline-2 | 15.89 (4.80)
  Change from Baseline-2 in Hyperactive/Impulsive Symptoms at Week 1 | -4.81 (4.74)
  Change from Baseline-2 in Hyperactive/Impulsive Symptoms at Week 2 | -6.38 (5.94)
  Change from Baseline-2 in Hyperactive/Impulsive Symptoms at Week 3 | -8.70 (5.81)
  Change from Baseline-2 in Hyperactive/Impulsive Symptoms at Week 4 | -9.00 (5.24)

7. Secondary Outcome: Change From Baseline-2 in the Clinical Global Impression of Severity (CGI-S) [ADHD Version] Scale Score
Description: CGI-S is an observer-rated scale that is used to assess the severity of the participants condition on a 7-point scale ranging from 1 to 7, where 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill. This rating is based upon observed and reported symptoms, behavior, and function in the past 7 days with a minimum score of 1 and maximum score of 7. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR. A negative change from Baseline indicates improvement.
Time Frame: Baseline-2, Weeks 1, 2, 3, 4 and 6 (Follow-up Visit)
Population: Per-protocol Population included all participants who met inclusion/exclusion criteria and completed the trial (4 weeks of drug treatment with evaluable data after Week 4) without major protocol violations. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  Baseline-2 | 4.68 (0.47)
  Change from Baseline-2 in CGI-S Score at Week 1 | -0.81 (0.70)
  Change from Baseline-2 in CGI-S Score at Week 2 | -1.30 (0.91)
  Change from Baseline-2 in CGI-S Score at Week 3 | -1.73 (0.96)
  Change from Baseline-2 in CGI-S Score at Week 4 | -1.89 (1.13)
  Change from Baseline-2 in CGI-S Score at Week 6 (Follow-up): number analyzed (Participants) | 36
  Change from Baseline-2 in CGI-S Score at Week 6 (Follow-up) | -0.92 (0.91)

8. Secondary Outcome: Change From Baseline-2 in the Clinical Global Impression of Improvement (CGl-I) [ADHD Version] Scale Score
Description: CGl-I is an observer-rated scale to assess how much the participant's illness has improved or worsened relative to a Baseline state, with scores ranging from 1 to 7. It consists of a 7-point scale ranging from 1 to 7, where 1=very much improved; 2=much improved; 3=minimally improved; 4=no change from Baseline-2 (the initiation of treatment); 5=minimally worse; 6=much worse; and 7=very much worse since the initiation of treatment. Improvement is defined as a score of 1=very much improved or 2=much improved on the scale. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR.
Time Frame: Baseline-2, Weeks 1, 2, 3, 4 and 6 (Follow-up)
Population: Data for this outcome measure was not collected as Baseline-2 CGI-I values were not recorded.
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Responders to the CGl-I (ADHD Version) Scale
Description: CGl-I is an observer-rated scale to assess how much the participant's illness has improved or worsened relative to a Baseline state, with scores ranging from 1 to 7. It consists of a 7-point scale ranging from 1 to 7, where 1=very much improved; 2=much improved; 3=minimally improved; 4=no change from Baseline-2 (the initiation of treatment); 5=minimally worse; 6=much worse; and 7=very much worse since the initiation of treatment. Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale. Responders are defined as those who had CGI-I (ADHD version) scores of much or very much improved.
Time Frame: Weeks 4 and 6 (Follow-up Visit)
Population: We have exhausted all efforts to locate this data and it has since been destroyed, therefore no data is available to report for this outcome measure.
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline-2 in the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a brief method of assessing both behavior and ideation that tracks all suicidal events, and provides a summary of suicidality. It assesses the lethality of attempts and other features of ideation (frequency, duration, controllability, reasons for ideation, and deterrents), all of which are significantly predictive of completed suicide. Severity of suicidal ideation is rated on a 6-point scale from 0=no ideation present to 5=active ideation with plan and intent. Suicidal behavior was collected as presence/absence of actual attempts, non-suicidal self-injurious behavior, interrupted attempts, aborted attempts, preparatory acts or behavior, and any suicidal behavior.
Time Frame: Baseline-2, Weeks 1, 4, and 6 (Follow-up Visit)
Population: as for outcome 9
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline-2 on the Profile of Mood States, Second Edition, Short Version 2A (POMS 2-A Short) at Week 4
Description: POMS 2-A Short version consists of a subset of 35 items from the full-length version of 72 mood adjectives assessing 7 mood domains namely, anger-hostility, confusion-bewilderment, depression-dejection, fatigue-inertia, tension-anxiety, vigor-activity, and friendliness. High scores indicate better vigor-activity and friendliness, but more severe symptoms for the five other domains. In addition, the Total Mood Disturbance (TMD) score is calculated from anger-hostility, confusion-bewilderment, depression-dejection, fatigue-inertia, tension-anxiety, and vigor-activity. Participants rated each of the 35 items using 4-point Likert-type scale (0=much unlike this; 3=much like this). Items from each domain are summed T-score such that total scores were in the negative-mood direction (i.e., higher scores indicate greater experience of negative moods). Total scores range from 0 to 100. TMD is calculated based on a standard value (mean of 50 and standard deviation of 10).
Time Frame: Baseline-2 and Week 4
Population: Per-protocol Population included all participants who met inclusion/exclusion criteria and completed the trial (4 weeks of drug treatment with evaluable data after Week 4) without major protocol violations. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR. Change from Baseline-2 for the POMS 2-A Short version scale is calculated using summary T-scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  TMD at Baseline-2 | 49.81 (8.34)
  Change from Baseline-2 in TMD at Week 4 | -2.81 (8.08)
  Tension-Anxiety at Baseline-2 | 48.65 (9.41)
  Change from Baseline-2 in Tension-Anxiety at Week 4 | -3.92 (8.38)
  Depression-Dejection at Baseline-2 | 45.41 (5.09)
  Change from Baseline-2 in Depression-Dejection at Week 4 | 0.05 (5.82)
  Anger-Hostility at Baseline-2 | 46.70 (7.07)
  Change from Baseline-2 in Anger-Hostility at Week 4 | -1.78 (5.52)
  Fatigue-Inertia at Baseline-2 | 44.62 (9.41)
  Change from Baseline-2 in Fatigue-Inertia at Week 4 | -1.73 (8.28)
  Confusion- Bewilderment at Baseline-2 | 54.54 (10.52)
  Change from Baseline-2 in Confusion-Bewilderment at Week 4 | -6.76 (10.20)
  Vigor-Activity at Baseline-2 | 53.95 (8.04)
  Change from Baseline-2 in Vigor-Activity at Week 4 | -3.16 (7.87)
  Friendliness at Baseline-2 | 50.59 (7.47)
  Change from Baseline-2 in Friendliness at Week 4 | -0.19 (7.05)

12. Secondary Outcome: Change From Baseline-2 on the Wender-Reimherr Adult Attention Deficit Disorder Scale (WRAADDS) at Week 4
Description: WRAADDS is used to measure the severity of symptoms in adults with ADHD. This structured interview consists of 28 items in 7 psychopathologic domains, which were rated by a clinical expert on a 0 to 2-point Likert scale. The psychopathologic 7 domains are inattention, hyperactivity, affective lability, hot temper, stress intolerance, disorganization, and impulsivity. The scale rated individual items from 0 to 2 (0=not present, 1=mild, 2=clearly present) and summarized each of the 7 categories on a 0-to-4 scale (0=none, 1=mild, 2=moderate, 3=quite a bit, 4=very much). The WRAADDS total score is defined as sum of all 28 item sub scores (range 0 to 56), higher scores indicate worsening of symptoms. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with CTN SR. A negative change from Baseline indicates improvement. Change from Baseline-2 for the WRAADDS scale is calculated using total scores.
Time Frame: Baseline-2 and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  WRAADDS Total Score at Baseline-2 | 33.59 (7.86)
  Change from Baseline-2 in WRAADDS Total Score at Week 4 | -15.59 (12.25)

13. Secondary Outcome: Change From Baseline-2 on the Weiss Functional Impairment Rating Scale - Self Report (WFIRS-S) at Week 4
Description: The WFIRS-S is a validated rating scale used to capture functional difficulties in the lives of individuals with ADHD. It investigates emotional or behavioral problems and is comprised of 69 items grouped into six domains: family (8 items), work (11 items), school (10 items, includes learning [4 items] and behavior [6 items]), life skills (12 items), self-concept (5 items), social (9 items), and risky (14 items). It uses a 4-point Likert scale where 0=never or not at all, 1=sometimes or somewhat, 2=often or much, and 3=very often or very much. Any item rating of 2 or 3 was considered in the clinically impaired range. A total score was derived by summing all scores from every domain, ranging from 0 to 207 with higher scores=greater ADHD-related functional impairment.
Time Frame: Baseline and Week 4
Population: Per-protocol Population included all participants who met inclusion/exclusion criteria and completed the trial (4 weeks of drug treatment with evaluable data after Week 4) without major protocol violations. Baseline-2 is defined as an end of 1-week SB placebo run-in and beginning of treatment with EB-1020 SR. A negative change from Baseline indicates improvement. Change from Baseline-2 for the WFIRS-S scale is calculated using average total scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 37
score on a scale
  WFIRS-S Total Score at Baseline-2 | 0.723 (0.304)
  Change from Baseline-2 in WFIRS-S Total Score at Week 4 | -0.258 (0.276)

14. Secondary Outcome: Change From Week 4 to End of Discontinuation Phase (Follow-up) on the ADHD-RS-IV
Description: The change on the ADHD-RS-IV was used to assess relapse of symptoms after end of investigational product administration.
Time Frame: Week 4 and end of Discontinuation Phase (Week 6)
Population: as for outcome 9
Arm/Group | Centanafadine SR 100-500 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline-2 through end of the study (Up to Week 6)
Description: Safety Population included all participants who received at least 1 dose of CTN SR (not placebo) as indicated in the treatment regimen.
Arm/Group | Centanafadine SR 100-500 mg
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 1/41
Other Adverse Events (participants affected / at risk) | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Centanafadine SR 100-500 mg (N=41)
Cerebrovascular accident (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Centanafadine SR 100-500 mg (N=41)
Tachycardia (Cardiac disorders) | 2
Diarrhea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 6
Headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 4
Irritability (Psychiatric disorders) | 4
Abnormal dreams (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 3
Middle insomnia (Psychiatric disorders) | 3
Lethargy (Psychiatric disorders) | 3
Dysphoria (Psychiatric disorders) | 3
Erectile dysfunction (Psychiatric disorders) | 2
Somnolence (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.